CLINICAL TRIAL: NCT02120664
Title: A Multicenter, Multicountry Study to Calibrate Florbetapir (18F) PET Imaging Data to the Centiloid Scale Based on 11C-PiB
Brief Title: Florbetapir Calibration to the Centiloid Scale
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A22
Record Dates: First submitted 2014-04-17; First posted 2014-04-23 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amyloid Negative Subjects (Experimental): Approximately 10 cognitively normal young subjects will receive a single i.v. bolus injection of approximately 370 megabecquerel (MBq) (10 millicurie [mCi]) florbetapir (18F) and a single i.v. bolus injection of approximately 555 MBq (15 mCi) 11C-PiB.
  Interventions: Drug: Florbetapir (18F); Drug: 11C-PiB
- Amyloid Positive Subjects (Experimental): Approximately 25 subjects with a range of amyloid density comprised of subjects clinically diagnosed with Alzheimer's Disease (AD) and subjects at risk for elevated amyloid density will receive a single i.v. bolus injection of approximately 370 MBq (10 mCi) florbetapir (18F) and a single i.v. bolus injection of approximately 555 MBq (15 mCi) 11C-PiB.
  Interventions: Drug: Florbetapir (18F); Drug: 11C-PiB

INTERVENTIONS:
Drug: Florbetapir (18F)
  Other Names: Florbetapir F 18; Amyvid; 18F-AV-45
Drug: 11C-PiB
  Other Names: Pittsburgh Compound B

SUMMARY:
This study is designed to demonstrate the conversion of florbetapir (18F) Positron Emission Tomography (PET) Standard Uptake Value ratio (SUVr) to Centiloid units.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively Normal Subjects

  * Males or females ≥ 21 and ≤ 45 years of age
  * Mini-mental state examination (MMSE) ≥ 29
* Clinically Diagnosed AD Subject

  * Males or females ≥ 50 years of age
  * Meet clinical criteria for dementia due to probable AD
  * MMSE ≥ 16 and ≤ 26
* Possible AD Subject

  * Males or females ≥ 50 years of age
  * Meet clinical criteria for dementia due to possible AD
  * MMSE ≥ 16 and ≤ 26
* MCI Subject

  * Males or females ≥ 60 years of age with cognitive impairment (not dementia)
  * MMSE >24 and <29
* At Risk Elderly Subject

  * Cognitively normal males or females that are known ApoE4 carriers and ≥ 75 years of age
  * MMSE ≥ 27

Exclusion Criteria:

* Have had or currently have a diagnosis of neurodegenerative disorders other than AD
* Have a current serious or unstable illness that could interfere with completion of the study
* Subject has a known brain lesion, pathology or traumatic brain injury
* Have received or participated in a trial with investigational medications in the past 30 days
* Have had a radiopharmaceutical imaging or treatment procedure within 7 days of study imaging session
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (2):
- Research Site, Pittsburgh, Pennsylvania, United States
- Research Site, Heidelberg, Victoria, Australia

REFERENCES:
- [Background] Klunk WE, Koeppe RA, Price JC, Benzinger TL, Devous MD Sr, Jagust WJ, Johnson KA, Mathis CA, Minhas D, Pontecorvo MJ, Rowe CC, Skovronsky DM, Mintun MA. The Centiloid Project: standardizing quantitative amyloid plaque estimation by PET. Alzheimers Dement. 2015 Jan;11(1):1-15.e1-4. doi: 10.1016/j.jalz.2014.07.003. Epub 2014 Oct 28. PMID 25443857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 14 April 2014; Last subject completed: 18 September 2015
Groups:
- Clincally Diagnosed AD: Patients meeting clinical criteria for dementia due to probable Alzheimer's Disease (AD)
- Possible AD: Patients meeting clinical criteria for dementia due to possible Alzheimer's Disease
- Mild Cognitive Impairment (MCI): Patients with a clinical diagnosis of Mild Cognitive Impairment (MCI) and not dementia. Age is 60 years or greater
- At Risk Elderly: Elderly patients, 75 years or older, who are known ApoE4 gene carriers, and cognitively normal
- Young Healthy Controls (YHC): Cognitively normal young subjects between 21 and 45 years of age (inclusive)
Period: Overall Study
Arm/Group | Clincally Diagnosed AD | Possible AD | Mild Cognitive Impairment (MCI) | At Risk Elderly | Young Healthy Controls (YHC)
Started | 10 | 4 | 7 | 4 | 10
Completed | 10 | 4 | 7 | 3 | 10
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects receiving at least one dose of florbetapir
Groups:
- Total: Total of all reporting groups
Arm/Group | Clincally Diagnosed AD | Possible AD | Mild Cognitive Impairment (MCI) | At Risk Elderly | Young Healthy Controls (YHC) | Total
Number analyzed (Participants) | 10 | 4 | 7 | 4 | 10 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (4.94) | 66 (4.76) | 79.9 (8.47) | 79.3 (2.5) | 27.3 (4.83) | 60.1 (22.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 0 | 7 | 15
  Male | 5 | 2 | 6 | 4 | 3 | 20
Mini Mental Status Exam [Mean (Standard Deviation); unit: units on a scale] — Mini Mental Status Exam (MMSE) is a brief instrument used to assess cognitive function in elderly patients. The instrument is divided into 2 sections. The first section measures orientation, memory, and attention. The maximum score for the first section is 21. The second section tests the ability of the patient to name objects, follow verbal and written commands, write a sentence, and copy figures. The maximum score for the second section is 9. The range for the total MMSE score is 0 to 30. Higher scores indicate higher cognitive function.
  units on a scale | 23.7 (2.45) | 21.8 (4.92) | 26.4 (1.27) | 29.3 (0.96) | 29.5 (0.53) | 26.3 (3.55)

OUTCOME MEASURES:

1. Primary Outcome: Florbetapir SUVr Conversion to Centiloid Units
Description: Conversion of florbetapir (18F) positron emission tomography (PET) standard uptake value ratio (SUVr) to Centiloid units. The Centiloid is anchored at values of 0 and 100 corresponding to the median Pittsburgh Compound B (11C-PiB) SUVr value for a representative group of young (<45) cognitively and medically healthy control subjects (YHC) and the median SUVr value for a representative group of 11C-PiB positive patients diagnosed with Alzheimer's disease, respectively. A cortical average to cerebellum SUVr was used for this outcome measure.
Time Frame: up to 70 minutes post injection
Population: All participants receiving both a florbetapir and a PiB scan per protocol. One subject in the possible AD group did not complete a florbetapir scan due to excessive movement. One subject in the at risk elderly group elected to leave the study before the second PET scan.
Measure: Mean (Standard Deviation); unit: centiloid
Arm/Group | Clincally Diagnosed AD | Possible AD | Mild Cognitive Impairment (MCI) | At Risk Elderly | Young Healthy Controls (YHC)
Number analyzed (Participants) | 10 | 3 | 7 | 3 | 10
centiloid | 82.44 (45.623) | 50.75 (60.383) | 81.19 (66.357) | 14.93 (35.885) | 5.24 (11.981)

2. Secondary Outcome: Correlation of Florbetapir (18F) Centiloid and 11C-PiB Centiloid
Description: Correlation coefficient between 11C-PiB and florbetapir (18F) SUVr as converted to centiloid units. The Centiloid is anchored at values of 0 and 100 corresponding to the median Pittsburgh Compound B (11C-PiB) SUVr value for a representative group of young (<45) cognitively and medically healthy control subjects (YHC) and the median SUVr value for a representative group of 11C-PiB positive patients diagnosed with Alzheimer's disease, respectively. A cortical average to cerebellum SUVr was used for this outcome measure.
Time Frame: up to 70 minutes post injection
Population: All participants receiving both a florbetapir and a PiB scan per protocol. One subject in the possible AD group did not complete the florbetapir scan due to excessive movement. One subject in the at risk elderly group elected to leave the study before the second PET scan.
Measure: Mean (Standard Deviation); unit: centiloid
Arm/Group | Clincally Diagnosed AD | Possible AD | Mild Cognitive Impairment (MCI) | At Risk Elderly | Young Healthy Controls (YHC)
Number analyzed (Participants) | 10 | 3 | 7 | 3 | 10
centiloid
  Florbetapir | 82.44 (45.623) | 50.75 (60.383) | 81.19 (66.357) | 14.93 (35.885) | 5.24 (11.981)
  11C-PiB | 87.18 (41.105) | 54.52 (56.511) | 74.33 (57.597) | 26.39 (37.464) | 0.73 (2.414)
Statistical Analysis 1: Comparison: Clincally Diagnosed AD vs Possible AD vs Mild Cognitive Impairment (MCI) vs At Risk Elderly vs Young Healthy Controls (YHC); Test type: Superiority or Other; Regression, Linear; R squared = 0.907

3. Secondary Outcome: Variability of PET Images in Young Healthy Control Subjects.
Description: Coefficient of variation for 11C-PiB and florbetapir (18F) SUVr. A cortical average to cerebellum SUVr was used for this outcome measure.
Time Frame: up to 70 minutes post injection
Population: Young healthy controls enrolled in the study
Measure: Mean (Standard Deviation); unit: SUVr
Groups:
- PiB SUVR Variability: Variability of standardized uptake value ratio (SUVR) for PiB scans in young healthy controls
- Florbetapir SUVR Variability: Variability of standardized uptake value ratio (SUVR) for florbetapir scans in young healthy controls
Arm/Group | PiB SUVR Variability | Florbetapir SUVR Variability
Number analyzed (Participants) | 10 | 10
SUVr | 1.01 (0.026) | 0.98 (0.066)
Statistical Analysis 1: Comparison: PiB SUVR Variability; Test type: Superiority or Other; Coefficient of Variation = 2.53
Statistical Analysis 2: Comparison: Florbetapir SUVR Variability; Test type: Superiority or Other; Coefficient of Variation = 6.69

ADVERSE EVENTS:
Time Frame: within 48 hours of scan as noted by group title
Groups:
- Florbetapir Only: Events occurring within 48 hours following florbetapir scans only
- PiB Only: Events occurring within 48 hours of PiB scans only
- Both: Events occurring within 48 hours of both florbetapir and PiB scans
- Total: Events following Florbetapir (florbetapir only and both)
Arm/Group | Florbetapir Only | PiB Only | Both | Total
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days